CLINICAL TRIAL: NCT01871337
Title: A Clinical Trial for the Efficacy of Paula Method ( Circular Muscle Exercise) in Women With Multiple Sclerosis Who Suffer From Urinary Incontinence
Brief Title: Exercises for Urinary Incontinence(UI) of Women With Multiple Sclerosis (MS)
Acronym: UI-MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UI_MS_HMO
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2012-12

CONDITIONS: Urinary Incontinence;; Multiple Sclerosis
Keywords: Multiple Sclerosis; urinary incontinence
MeSH Terms: conditions — Urinary Incontinence; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paula method (Experimental): the Paula method, a circular muscle exercise, invented in Israel by Paula Garbourg.The method is based on the principle that all sphincters in the body are synchronized, with the movement of one affecting the other.One can rehabilitate damaged muscles by contracting and relaxing specific "circular" muscles in other parts of the body.
  Interventions: Behavioral: Paula method

INTERVENTIONS:
Behavioral: Paula method — The Paula method will be taught to the participants by several registered Paula instructors. Subjects allocated to this intervention will receive one 45-minute group session per week for 12 weeks (with up to 30 minutes for personal questions regarding the exercises). This length of time is crucial because it has been demonstrated that it take three months for women to adequately learn the exercises in order for them to practice independently at home. Participants will be encouraged to practice daily for 15 minutes and report their at- home training.
  Other Names: Circular muscle exercises

SUMMARY:
This study will examine whether the Paula method is an effective treatment for UI and the correlating LUTD symptoms. We assume that the Paula method, a simple, non-aerobic exercise method that significantly decreased urinary incontinence in women with MIX in two randomized controlled trials, would also be effective in Multiple Sclerosis (MS) patients with UI. The secondary aim is to evaluate the effectiveness in terms of MS general physical functioning, quality of life and sexual function and to detect adherence and continuity six months post intervention.

DETAILED DESCRIPTION:
The patient will be examined by the neurologist at the MS clinic, at the Hadassah University Medical Center. Patients who meet the inclusion criteria will receive an explanation, and will sign informed consent. She will be asked to complete the baseline questionnaires. Than the patient will be assigned to an exercise group. After 12 weeks the patient will be asked to complete post intervention questionnaire. Apart from the weekly lesson, women will be asked to exercise at home for 15 minutes a day. After six months she will be invited again for a neurological examination and filling an additional questionnaire.

ELIGIBILITY:
Inclusion Criteria:

women ≥18 years old; who have complained of urine leakage in the past four weeks; MS diagnosed with an Expanded Disability Status Scale (EDSS)≤7.5; literate in Hebrew and/or English; suffering from UI at least in the 4 last weeks prior to recruitment

Exclusion Criteria:

pregnant or breastfeeding women, those within 12 weeks of delivery; 6 weeks of abortion; six months of pelvic surgery; symptomatic urinary tract infection (UTI); more than grade 2 genital prolapse, permanent catheterization for urination; women taking medications for UI less then 3 months and women who exercise on regular basis in Paula method.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Urinary Incontinence ,measured by The ICIQ-SF Short Form questionnaire | two years

SECONDARY OUTCOMES:
quality of life, sexual function and mobility | two years
  Questionnaire for Urinary Incontinence Diagnosis (QUID); The Incontinence Quality of Life Questionnaire (I -QOL); The Pelvic Organ Prolapse/ Urinary Incontinence Sexual Questionnaire (PISQ-12); Expanded Disability Status Scale (EDSS);Demographic data questionnaire, General health and Paula Method Evaluation; Long term (6 months after the end of the intervention) questionnaire;

CONTACTS AND LOCATIONS:
Overall Officials: Adi Vaknin, MD, Principal Investigator — Hadassah University Hospital
Locations (2):
- Israel (2):
  - Hadassah University Hospital, Jerusalem
  - Hadassah Hospital, Jerusalem